CLINICAL TRIAL: NCT05300009
Title: Efficacy and Safety of Topical Methotrexate Gel 1% Coupled With Microneedling in Treatment of Warts : A Prospective Controlled Randomized Trial
Brief Title: Efficacy and Safety of Topical Methotrexate Gel 1% Coupled With Microneedling in Treatment of Warts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khulood Fadhl Ahmed Alhakami, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MGMW
Record Dates: First submitted 2022-03-04; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Warts
MeSH Terms: conditions — Warts | interventions — Family Characteristics; Percutaneous Collagen Induction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- topical methotrexate hydrogel 1% coupled with microneedling (Experimental): patients who will receive topical methotrexate hydrogel 1% coupled with microneedling
  Interventions: Combination Product: topical methotrexate hydrogel 1% coupled with microneedling.
- cryotherapy (Active Comparator): patients who will receive cryotherapy
  Interventions: Other: Liquid nitrogen

INTERVENTIONS:
Combination Product: topical methotrexate hydrogel 1% coupled with microneedling. — Microneedling will be performed on each wart for a maximum 5 lesions per patient using dermapen (Ostar rechargeable dermapen, OB-DG 03N, Ostar Beauty Sci-Tech Co, Beijing, China) supplied with 12 needles arranged in rows. The penetration depth was adjusted at 2-mm, endpoint was pinpoint bleeding and the dermapen will be held by the hand in a vertical direction on the wart. Then topical methotrexate 1% gel will be applied on the lesions every session.
  Arms: topical methotrexate hydrogel 1% coupled with microneedling
Other: Liquid nitrogen — The wart is frozen for 10 to 30 seconds until a 1- to 2-mm ice ball halo surrounds the targeted area.
  The sessions were performed every 2 week until complete clearance for a maximum of six sessions.
  Arms: cryotherapy

SUMMARY:
To study the clinical efficacy of the topically applied MTX hydrogel preparation combined with microneedling to increase drug delivery and efficacy in comparison with cryotherapy in treatment of warts.

DETAILED DESCRIPTION:
Warts are benign proliferation of skin and mucosa caused by the human papilloma virus (HPV). Currently, over 170 HPV types have been identified. Certain HPV types tend to infect skin at anatomical sites, for an example, palmoplantar warts are usually caused by Serotypes 1, 2, and 4; however, warts of any HPV type may occur at any site. Warts are transmitted by direct or indirect contact, and predisposing factors include disruption to the normal epithelial barrier.

There are several modalities for treatment of warts including cryotherapy, electrocoagulation, topical salicylic acid, topical 5-fluorouracil, and laser surgery. All these treatment options can be painful, time-consuming, and/or expensive, and none is considered the gold standard.

Treatments for warts have also included intralesional injections of tuberculin purified protein derivative (PPD), measles, mumps, and rubella vaccine (MMR), and Candida albicans antigen (candidin). This treatment approach is known as intralesional immunotherapy as it is thought that these modalities activate the immune system to recognize the virus, leading to wart clearance

. MTX as an antimetabolite and antifolate drug is a time-tested effective treatment extensively used orally or parenteral in various autoimmune disorders like psoriasis, psoriatic arthritis, alopecia areata, lupus erythematosus, and rheumatoid arthritis in low to moderate doses with good efficacy, safety, and tolerability on a long-term basis

MTX is appropriate for rapidly growing tumors since it inhibits DNA synthesis in actively dividing cells. MTX is a folic acid analog that binds to the dihydrofolate reductase, blocking the formation of tetrahydrofolate and preventing the synthesis of the purine nucleotide thymidine .

Antiviral effect of MTX was observed in the treatment of Zika virus infected cells explaining the antiviral effect of MTX through inhibition of dihydrofolate reductase ..

A literature review shows that intralesional MTX has been successfully used for several indications with no complications reported.

Unlike systemic MXT, topical preparations of the drug, that was adapted for the treatment of localized lesions, showed nonsignificant related hepatotoxic and hematologic adverse effects .

Previous studies used intralesional MTX injection in the treatment of viral warts with different concentrations and revealed that intralesional MTX was less effective in treating plantar warts .

Since MTX is used for various diseases via different routes of administration, the development of novel drug delivery systems to improve its pharmacokinetic properties and targetability is a necessary step for future investigations .

Controlling the burst release and the introduction of new routes of administration would be possible if the drug could be formulated using different delivery systems. Among various drug delivery systems proposed for MTX delivery, great attention has been directed to hydrogels due to their unique and attractive characteristics .

Microneedling is a fine needle that penetrates the skin to induce micro-injuries leading to production of collagen fibers and release of growth factors .

Microneedling has been used as an adjuvant therapy helping a drug delivery and also used in treatment of various dermatologic diseases .

In this study, the investigators chose the hydrogel formulation at a concentration of 1%w/v as a topical MTX form coupled with microneedling to increase the efficacy of methotrexate in treatment of warts. Hydrogel used will be optimized for biocompatibility, consistency and chemical compatibility with methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years up to 60 years old.
* Patients with plantar or common warts.

Exclusion Criteria:

* pregnancy and lactation
* immunosuppression or being under any kind of treatment causing absolute or relative immunosuppression.
* history of any bleeding, clotting disorder or using anticoagulants.
* chronic systemic diseases such as chronic renal failure, hepatic insufficiency, and cardiovascular disorders.
* concurrent use of systemic or topical treatments of warts .

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Complete resolution of all treated wart(s). | 8 weeks
  Proportion of participants with total remission of wart(s) at the end of the intervention in the two arms of the clinical trial assessed by the investigator and photographic evaluation .
  Complete response: responders who show 100% improvement (disappearance of all warts and return to normal skin markings).
Partial resolution | 8 weeks
  Number of subjects achieving partial resolution of treated wart(s) at the end of the intervention in the two arms of the clinical trial assessed by the investigator, photographic evaluation and The following grading system :
  Marked response: responders who show 76 to 99% decrease in number and/or decrease in apparent size, as assessed by a clinician and photographic evaluation also known as near-complete response.
  Moderate response: partial responders show 25 to 75% improvement. No or minimal response: less than 25% decrease in size/numbers of all warts. the stud
Incidence of adverse events | 8 weeks
  Proportion of participants that developed a serious side effect in the two arms during the clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Khulood F Alhakami, M.B.B.CH, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghittoni R, Accardi R, Chiocca S, Tommasino M. Role of human papillomaviruses in carcinogenesis. Ecancermedicalscience. 2015 Apr 29;9:526. doi: 10.3332/ecancer.2015.526. eCollection 2015. PMID 25987895
- [Background] Kimura U, Takeuchi K, Kinoshita A, Takamori K, Suga Y. Long-pulsed 1064-nm neodymium:yttrium-aluminum-garnet laser treatment for refractory warts on hands and feet. J Dermatol. 2014 Mar;41(3):252-7. doi: 10.1111/1346-8138.12411. Epub 2014 Feb 10. PMID 24506821
- [Background] Shaheen MA, Salem SA, Fouad DA, El-Fatah AA. Intralesional tuberculin (PPD) versus measles, mumps, rubella (MMR) vaccine in treatment of multiple warts: a comparative clinical and immunological study. Dermatol Ther. 2015 Jul-Aug;28(4):194-200. doi: 10.1111/dth.12230. Epub 2015 Apr 6. PMID 25847793
- [Background] Sung JY, Hong JH, Kang HS, Choi I, Lim SD, Lee JK, Seok JH, Lee JH, Hur GM. Methotrexate suppresses the interleukin-6 induced generation of reactive oxygen species in the synoviocytes of rheumatoid arthritis. Immunopharmacology. 2000 Apr;47(1):35-44. doi: 10.1016/s0162-3109(99)00185-x. PMID 10708808
- [Background] Cipriani P, Ruscitti P, Carubbi F, Liakouli V, Giacomelli R. Methotrexate: an old new drug in autoimmune disease. Expert Rev Clin Immunol. 2014 Nov;10(11):1519-30. doi: 10.1586/1744666X.2014.962996. Epub 2014 Sep 22. PMID 25245537
- [Background] Beck S, Zhu Z, Oliveira MF, Smith DM, Rich JN, Bernatchez JA, Siqueira-Neto JL. Mechanism of Action of Methotrexate Against Zika Virus. Viruses. 2019 Apr 10;11(4):338. doi: 10.3390/v11040338. PMID 30974762
- [Background] Duarte AA, Carneiro GP, Murari CM, Jesus LCB. Nail psoriasis treated with intralesional methotrexate infiltration. An Bras Dermatol. 2019 Oct 17;94(4):491-492. doi: 10.1590/abd1806-4841.20198170. eCollection 2019. No abstract available. PMID 31644634
- [Background] Sutton L, Swinehart JM, Cato A, Kaplan AS. A clinical study to determine the efficacy and safety of 1% methotrexate/Azone (MAZ) gel applied topically once daily in patients with psoriasis vulgaris. Int J Dermatol. 2001 Jul;40(7):464-7. doi: 10.1046/j.1365-4362.2001.01244.x. No abstract available. PMID 11679005
- [Background] Abdo HM, Elrewiny EM, Elkholy MS, Ibrahim SM. Efficacy of intralesional methotrexate in the treatment of plantar warts. Dermatol Ther. 2020 Mar;33(2):e13228. doi: 10.1111/dth.13228. Epub 2020 Jan 29. PMID 31965678
- [Background] Dehshahri A, Kumar A, Madamsetty VS, Uzieliene I, Tavakol S, Azedi F, Fekri HS, Zarrabi A, Mohammadinejad R, Thakur VK. New Horizons in Hydrogels for Methotrexate Delivery. Gels. 2020 Dec 30;7(1):2. doi: 10.3390/gels7010002. PMID 33396629
- [Background] Badran MM, Kuntsche J, Fahr A. Skin penetration enhancement by a microneedle device (Dermaroller) in vitro: dependency on needle size and applied formulation. Eur J Pharm Sci. 2009 Mar 2;36(4-5):511-23. doi: 10.1016/j.ejps.2008.12.008. Epub 2008 Dec 25. PMID 19146954
- [Background] Ita K. Dissolving microneedles for transdermal drug delivery: Advances and challenges. Biomed Pharmacother. 2017 Sep;93:1116-1127. doi: 10.1016/j.biopha.2017.07.019. Epub 2017 Jul 19. PMID 28738520